CLINICAL TRIAL: NCT02061007
Title: Biomarker Correlates of Hypoxia in Metastatic Melanoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no accrual
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MCC-17034
Record Dates: First submitted 2014-02-10; First posted 2014-02-12 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Melanoma; Skin Cancer
Keywords: skin cancer
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — pimonidazole; fluoromisonidazole; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Scans, Surgery and Follow-up (Experimental): Pre-surgery scans, surgical resection and post-surgery follow-up. All patients will receive a fluorodeoxyglucose (FDG)-PET scan as part of standard of care. This scan must be completed within 28 days of surgery for the patient to be eligible. All patients will be offered the opportunity to receive an additional 18F-FMISO-PET scan, until 18 such scans are administered. Prior to surgery, patients will be administered a single dose of 0.5 g/m^2 (approximately 13 mg/kg) of oral Hypoxyprobe™-1 (pimonidazole, HCl).
  Interventions: Drug: Pimonidazole hydrochloride (Hypoxyprobe™-1); Drug: Optional 18F-FMISO PET scan (18F-fluoromisonidazole); Procedure: Surgical Resection of Melanoma Metastases

INTERVENTIONS:
Drug: Pimonidazole hydrochloride (Hypoxyprobe™-1) — Prior to surgery, patients will be administered a single dose of 0.5 g/m^2 (approximately 13 mg/kg) of oral Hypoxyprobe™-1 (pimonidazole, HCl).
  Other Names: Hypoxyprobe™-1; pimonidazole; HCI; pimo
Drug: Optional 18F-FMISO PET scan (18F-fluoromisonidazole) — All patients will be offered the opportunity to receive an additional 18F-FMISO-PET scan, until 18 such scans are administered.
  Other Names: 18F-fluoromisonidazole; 18F-MISO
Procedure: Surgical Resection of Melanoma Metastases — Participants will undergo surgical resection of melanoma metastases within 16 - 24 hours of consuming oral pimonidazole. Pimonidazole staining will be done on formalin-fixed and paraffin-embedded (FFPE) tissues for pimonidazole analysis. All participants will be contacted 24-72 hours post-surgery to be assessed for any adverse events (AEs) related to surgery, pimonidazole consumption and 18F-FMISO (when applicable).
  Other Names: surgery; resection

SUMMARY:
The purpose of this study is to determine if magnetic resonance imaging (MRI) or positron emission tomography (PET) imaging can be used to help doctors determine how much oxygen a tumor is getting. Hypoxyprobe will be used to determine the levels of oxygen post-surgery in the current study. If the study is successful, then imaging can be used to determine a tumor's oxygen status even in patients who are not getting surgery.

Investigators want to find out how much oxygen is in the participants tumor based on how much pimo is present, and correlate this with the results of their MRI and 18F-fluoromisonidazole (FMISO) PET scan.

This study is also testing the investigational radioactive substance known as FMISO. FMISO is used during PET scans to help doctors see how much oxygen a tumor is getting. Participants might be asked to participate in an optional PET scan using FMISO.

DETAILED DESCRIPTION:
A pilot phase II imaging study to determine hypoxia in melanoma.

About 16 - 24 hours before surgery, participants will be asked to come to the study center to take the investigational agent oral pimonidazole (pimo) by mouth. Pimo is a substance that is able to enter tissue when there are low levels of oxygen present (hypoxia). When the tissue is removed and visualized under a microscope, the amount of pimo present is related to the amount of oxygen in that part of the tissue. The dose of pimo given to the participant will depend on their weight (13 mg pimo/kg body weight).

After surgery, a sample of the participant's tumor tissue will be viewed by doctors under a microscope to determine the amount of pimo present.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years or older with a histological diagnosis of locally advanced, recurrent or metastatic melanoma and be scheduled for clinically indicated surgical removal of one or more melanoma tumors. Additionally, patients must have a resectable tumor nodule ≥1 cm^3 (i.e., either a spherical tumor at least 1.0 cm in diameter or a tumor measuring at least 1x1x1 cm). Prior biopsy is not required for study participation.
* Not pregnant or nursing (as confirmed by serum pregnancy test if the patient is a woman of child-bearing potential). Participants must agree with use birth control for 30 days following pimonidazole administration.
* Adequate kidney and liver function as assessed by laboratory studies
* Must be able to undergo magnetic resonance imaging (MRI) scans
* Capable of providing informed consent and demonstrate a willingness to comply with all the study procedures and visits
* Eastern Cooperative Oncology Group (ECOG) score of 0 -1

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Patients who are contraindicated for MRI or gadolinium contrast agents due to:

  * Presence of metallic objects or implanted medical devices in body (i.e., cardiac pacemaker, aneurysm clips, surgical clips, prostheses, skin staples, implanted prostheses, artificial heart valves with steel parts, metal fragments, shrapnel, or other metal implants that would contraindicate MRI)
  * Sickle cell disease
  * Renal failure with estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m^2 based upon serum creatinine
  * Weight greater than 350 lbs (the weight limit for the MRI)
* Patients with known, active (i.e. not adequately treated with curative intent) malignancies other than melanoma
* Presence of any other co-existing condition which, in the judgment of the investigator, might increase the risk to the participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Percentage of Positive Biomarker Staining by Applicable Area | 6 weeks per participant
  Relationship between MRI and/or FMISO-PET imaging features and pimonidazole staining by immunohistochemical analysis in melanoma metastases. Investigators expect that the correlation between them is at least 0.45. With a 5% significance level, a total of 36 participants will provide 81% power to test a null hypothesis correlation of 0 versus an alternative hypothesis correlation of 0.45 using a two-sided test.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Zager, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute